CLINICAL TRIAL: NCT02033005
Title: Newborn Feeding and Infant Phenotype
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRO1461
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Breast Feeding
Keywords: Body Composition; Adipose Tissue; Intrahepatocellular Lipid; Infant; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Stool Breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Breastfed infants: >80% of feeds consisting of breast milk at both scanning points
- Formula-fed infants: >80% of feeds consisting of formula milk at both scanning points
- Mixed-fed infants: 20%-80% of feeds consisting of breast milk.

SUMMARY:
Breast feeding is believed to be beneficial to long-term health but how these effects are mediated is unknown. I suggest that this may be through effects on body composition and metabolism.

I will compare adipose tissue and liver fat deposition in healthy, full term breast and formula fed infants babies shortly after birth and around 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy baby
* Term baby
* Appropriate weight for gestational age (UK - WHO 2009 growth charts)

Exclusion Criteria:

* Infants of diabetic mothers
* Infants of smokers
* Infants fed non-commercial or non-cows milk based infant formulae

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy, full term, appropriate weight for gestational age infants recruited on the postnatal ward at Chelsea and Westminster Hospital, London, UK.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neena Modi, MBBS, MD, Principal Investigator — Imperial College London
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Gale C, Thomas EL, Jeffries S, Durighel G, Logan KM, Parkinson JR, Uthaya S, Santhakumaran S, Bell JD, Modi N. Adiposity and hepatic lipid in healthy full-term, breastfed, and formula-fed human infants: a prospective short-term longitudinal cohort study. Am J Clin Nutr. 2014 May;99(5):1034-40. doi: 10.3945/ajcn.113.080200. Epub 2014 Feb 26. PMID 24572562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants consisted of healthy, full term, appropriate weight-for-gestational age infants from 2 cohorts: recruited between November 1999 and October 2001 at the Hammersmith Hospital, and between March 2010 and May 2012 from the postnatal ward at Chelsea and Westminster Hospital.
Period: Overall Study
Arm/Group | Breastfed Infants | Mixed-fed Infants | Formula-fed Infants
Started | 80 | 9 | 35
Completed | 36 | 9 | 25
Not Completed | 44 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breastfed Infants | Mixed-fed Infants | Formula-fed Infants | Total
Number analyzed (Participants) | 36 | 9 | 25 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 9 | 25 | 70
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Days] | 13 [9 to 18] | 2 [1 to 10] | 16 [9 to 20] | 13 [9 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15 | 30
  Male | 25 | 5 | 10 | 40
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36 | 9 | 25 | 70
Weight [Mean (Standard Deviation); unit: kg] | 3.647 (0.421) | 3.332 (0.478) | 3.622 (0.595) | 3.598 (0.500)
Length [Mean (Standard Deviation); unit: m] | 0.533 (0.023) | 0.510 (0.025) | 0.523 (0.025) | 0.527 (0.025)
Head circumference [Mean (Standard Deviation); unit: cm] | 36.5 (1.4) | 35.0 (1.7) | 36 (1.6) | 36.1 (1.6)
Total adipose tissue [Median (Inter-Quartile Range); unit: l] | 0.710 [0.632 to 0.899] | 0.802 [0.620 to 0.949] | 0.722 [0.613 to 0.913] | 0.718 [0.621 to 0.921]
Total adipose tissue mass % [Median (Inter-Quartile Range); unit: Percentage of mass] | 17.5 [16.3 to 19.8] | 21.3 [18.9 to 22.1] | 18.3 [16.6 to 21.7] | 18.1 [16.4 to 21.5]
Superficial subcutaneous abdominal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.098 [0.077 to 0.122] | 0.110 [0.090 to 0.116] | 0.103 [0.075 to 0.14] | 0.101 [0.077 to 0.129]
Superficial subcutaneous non-abdominal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.512 [0.454 to 0.680] | 0.572 [0.423 to 0.692] | 0.521 [0.452 to 0.648] | 0.512 [0.446 to 0.669]
Deep subcutaneous abdominal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.015 [0.011 to 0.021] | 0.013 [0.011 to 0.024] | 0.019 [0.011 to 0.022] | 0.016 [0.011 to 0.022]
Deep subcutaneous non-abdominal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.012 [0.009 to 0.015] | 0.012 [0.012 to 0.014] | 0.013 [0.011 to 0.016] | 0.013 [0.010 to 0.015]
Internal abdominal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.017 [0.013 to 0.022] | 0.022 [0.014 to 0.027] | 0.017 [0.012 to 0.022] | 0.017 [0.013 to 0.023]
Internal non-abdominal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.054 [0.044 to 0.065] | 0.061 [0.051 to 0.078] | 0.052 [0.047 to 0.072] | 0.054 [0.045 to 0.070]
Total subcutaneous adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.633 [0.570 to 0.833] | 0.718 [0.484 to 0.950] | 0.654 [0.529 to 0.832] | 0.644 [0.553 to 0.835]
Total internal adipose tissue [Median (Inter-Quartile Range); unit: Litres] | 0.070 [0.056 to 0.086] | 0.084 [0.059 to 0.106] | 0.069 [0.055 to 0.091] | 0.070 [0.056 to 0.093]
Intrahepatocellular lipid [Median (Inter-Quartile Range); unit: Ratio of CH2 (methylene) to H2O (water)] | 0.662 [0.353 to 1.965] | 1.126 [0.695 to 1.573] | 1.197 [0.710 to 1.650] | 0.949 [0.521 to 1.711]

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Adipose Tissue Volume
Description: Difference in total adipose tissue volume, measured using whole body magnetic resonance imaging.
Time Frame: Between birth and 6-12 weeks age
Population: Reduced participant number for this analysis represents missing data for some infants at one scan point
Measure: Median (Inter-Quartile Range); unit: Litres
Groups:
- Breastfed: >80% of feeds consisting of breastmilk at both scanning points
Arm/Group | Breastfed | Mixed-fed Infants | Formula-fed Infants
Number analyzed (Participants) | 35 | 9 | 24
Litres | 0.718 [0.508 to 0.938] | 0.901 [0.452 to 1.053] | 0.775 [0.532 to 0.971]

2. Secondary Outcome: Change in Regional Adipose Tissue Distribution Compared to Breastfed Infants.
Description: Change in regional adipose tissue distribution (ratio of internal abdominal to total subcutaneous abdominal adipose tissue) measured using whole body magnetic resonance imaging
Time Frame: Between birth and 6-12 weeks age
Population: Reduced participant number for this analysis represents missing data for some infants at one scan point
Measure: Median (Inter-Quartile Range); unit: no unit (ratio)
Groups:
- Breastfed Infants: >80% of feeds consisting of breastmilk at both scanning points
Arm/Group | Breastfed Infants | Mixed-fed Infants | Formula-fed Infants
Number analyzed (Participants) | 35 | 9 | 24
no unit (ratio) | -0.07 [-0.09 to -0.02] | -0.06 [-0.08 to -0.02] | -0.03 [-0.07 to 0.01]

3. Secondary Outcome: Change in Intrahepatocellular Lipid Compared to Breastfed Infants.
Description: Change in intrahepatocellular lipid (IHCL) compared to breastfed infants, measured using in-vivo hepatic magnetic resonance spectroscopy
Time Frame: Between birth and 6-12 weeks age
Population: Reduced number of participants due to missing intrahepatocellular lipid data in some cases
Measure: Median (Inter-Quartile Range); unit: ratio of CH2 to water
Arm/Group | Breastfed Infants | Mixed-fed Infants | Formula-fed Infants
Number analyzed (Participants) | 30 | 4 | 20
ratio of CH2 to water | 1.192 [0.226 to 1.967] | -0.054 [-.672 to 1.837] | 1.095 [-0.280 to 1.746]

ADVERSE EVENTS:
Time Frame: 2 years and 2 months
Arm/Group | Breastfed Infants | Mixed-fed Infants | Formula-fed Infants
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/9 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/9 | 0/25
Other Adverse Events (participants affected / at risk) | 0/36 | 0/9 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes